CLINICAL TRIAL: NCT02769286
Title: Phase II Trial of AZD9291 in First Line Treatment of Lung Cancer Harboring Activating EGFR Mutation From Circulating Tumor DNA and Second Line Treatment After Acquired Resistance With T790M Mutation Detected From Circulating Tumor DNA
Brief Title: Osimertinib in First and Second Line Treatment of NSCLC Harboring EGFR Mutations From Circulating Tumor DNA
Acronym: LiquidLung-O
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-11075
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms; EGFR Gene Mutations
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osimertinib in cohort 1 (Experimental): Treatment efficacy of osimertinib will be assessed in patients with lung cancer harboring EGFR mutations which were detected from circulating tumor DNA
  Interventions: Drug: Osimertinib
- Osimertinib in cohort 2 (Experimental): Treatment efficacy of osimertinib will be assessed in patients with lung cancer harboring T790M which were detected from circulating tumor DNA
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Treatment efficacy of osimertinib will be assessed in patients with lung cancer harboring EGFR mutations (cohort 1) and those harboring T790M (cohort 2) which were detected from circulating tumor DNA
  Other Names: AZD9291

SUMMARY:
Treatment efficacy of osimertinib will be assessed in patients with lung cancer harboring activating epidermal growth factor receptor (EGFR) mutations (cohort 1) and those harboring T790M (cohort 2) which were detected from circulating tumor DNA

DETAILED DESCRIPTION:
This is a phase II, open-label, single centre study of AZD9291 administered orally in patients with advanced lung cancer with activating mutations of EGFR gene with or without T790M which were detected from circulating tumor DNA. EGFR-TKI naïve patients with activating EGFR mutation will be enrolled in cohort 1. Patients with acquired resistance to prior EGFR tyrosine kinase inhibitor (TKI) due to T790M mutation is going to be enrolled in cohort 2.

ELIGIBILITY:
Inclusion Criteria:

< Cohort 1 >

1. Provision of informed consent prior to any study specific procedures
2. Patients (male/female) must be > 18 years of age.
3. Locally advanced or metastatic non-small cell lung cancer, not amenable to curative surgery or radiotherapy with or without pathologic diagnosis
4. No prior exposure to EGFR TKI (multiple lines of prior cytotoxic chemotherapy are permitted.)
5. Activating EGFR mutation (G719X, exon 19 deletion, L858R, L861Q) detected from circulating tumor DNA either by PANA mutyper® or Cobas® EGFR mutation test.
6. Activating EGFR mutation (G719X, exon 19 deletion, L858R, L861Q) detected from tumor tissue or cytology specimen.
7. World Health Organization (WHO) performance status 0-2.
8. Patients must have a life expectancy ≥ 12 weeks.
9. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
10. Male patients should be willing to use barrier contraception.
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT)

< Cohort 2 >

1. Provision of informed consent prior to any study specific procedures
2. Patients (male/female) must be > 18 years of age.
3. Locally advanced or metastatic non-small cell lung cancer, not amenable to curative surgery or radiotherapy with or without pathologic diagnosis
4. Progression after prior exposure to gefitinib, erlotinib, afatinib or dacomitinib. Multiple lines of prior cytotoxic chemotherapy are permitted and there is no specified order of treatment.
5. Patients must fulfil one of the following:

   5.1) Activating EGFR mutation (G719X, exon 19 deletion, L858R, L861Q) from tumor tissue or cytology or circulating tumor DNA 5.2) Must have experienced clinical benefit from prior EGFR-TKI, according to the Jackman criteria (Jackman 2010) followed by systemic objective progression (RECIST) while on continuous treatment with EGFR-TKI
6. T790M mutation detected from circulating tumor DNA either by PANA mutyper® or Cobas® EGFR mutation test.
7. World Health Organization (WHO) performance status 0-2.
8. Patients must have a life expectancy ≥ 12 weeks.
9. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
10. Male patients should be willing to use barrier contraception.
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT)

Exclusion Criteria:

1. Previous treatment with AZD9291, or other 3rd generation EGFR TKI
2. Treatment with an investigational drug within five half-lives of the compound
3. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior) (Appendix A). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
4. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
6. Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable
7. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
8. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   Absolute neutrophil count <1.5 x 109/L Platelet count <100 x 109/L Haemoglobin <90 g/L Alanine aminotransferase >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
9. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9291
11. History of hypersensitivity to AZD9291 (or drugs with a similar chemical structure or class to AZD9291) or any excipients of these agents
12. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
13. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
14. Previous allogeneic bone marrow transplant.
15. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 2 months
  RECIST v1.1

SECONDARY OUTCOMES:
Sensitivity of testing methods | 2 weeks
  Percentage of positive cases among cases tested with Mutyper or Cobas
Progression free survival | 2 years
Duration of response | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Jackman D, Pao W, Riely GJ, Engelman JA, Kris MG, Janne PA, Lynch T, Johnson BE, Miller VA. Clinical definition of acquired resistance to epidermal growth factor receptor tyrosine kinase inhibitors in non-small-cell lung cancer. J Clin Oncol. 2010 Jan 10;28(2):357-60. doi: 10.1200/JCO.2009.24.7049. Epub 2009 Nov 30. PMID 19949011